CLINICAL TRIAL: NCT01562743
Title: An Open-label Long-term Extension Trial From Late Phase II of SPM 962 (243-07-003) in Patients With Restless Legs Syndrome
Brief Title: A Long-Term Extension Trial From Late Phase II of SPM 962 in Patients With Restless Legs Syndrome
Acronym: RLS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 243-07-004
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Idiopathic Restless Legs Syndrome
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPM 962 (Experimental): Rotigotine transdermal patch
  Interventions: Drug: SPM 962

INTERVENTIONS:
Drug: SPM 962 — Tansdermal patch
  Other Names: rotigotine

SUMMARY:
The aims of the trial are to assess the safety and the efficacy of SPM 962 following once-a-daily transdermal administration within a range of 2.25 to 6.75 mg/day in Japanese patients with restless legs syndrome (RLS) in a multi-center, open-label trial. The maximum treatment period is 53 weeks. The trial is an extension trial from the precedent 6-week, double-blind, randomized, placebo-controlled, parallel-group comparative trial(243-07-003). The trial is also for an exploratory investigation of incidence of augmentation, the most problematic complications in dopaminergic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the preceding trial 243-07-003 (NCT00666965)

Exclusion Criteria:

* Subject discontinued from the preceding trial 243-07-003 (NCT00666965)
* Subject had a serious adverse event which association with the investigational drug is not ruled out during trial 243-07-003
* Subject had a persistent serious adverse event at the baseline, which was observed and association with the investigational drug is ruled out during trial 243-07-003.
* Subject had persistent hallucination or delusion during trial 243-07-003.
* Subject had psychiatric conditions such as confusion, excitation, delirium, abnormal behaviour at the baseline.
* Subject had orthostatic hypotension or a systolic blood pressure (SBP) ≤ 100 mmHg and had a decrease of SBP from spine to standing position ≥ 30 mmHg at baseline.
* Subject had a history of epilepsy, convulsion etc. during trial 243-07-003.
* Subject developed serious ECG abnormality at the baseline.
* Subject had QTc-interval ≥ 500 msec at the baseline or subject had an increase of QTc-interval ≥ 60 msec from the baseline in the trial 243-07-003 and had a QTc-interval > 470 msec in female or > 450 msec in male at the baseline.
* Subject had a serum potassium level < 3.5 mEq/L at the end of the taper period in trial 243-07-003.
* Subject had a total bilirubin ≥ 3.0 mg/dL or AST(GOT) or ALT(GPT) greater than 2.5 times of the upper limit of the reference range (or ≥ 100 IU/L) at the end of the period in trial 243-07-003.
* Subject had BUN ≥ 30 mg/dL or serum creatinine ≥ 2.0 mg/dl at the end of the taper period in trial 243-07-003.
* Subject who planned pregnancy during the trial.
* Subject was judged to be inappropriate for this trial by the investigator for the reasons other than above.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

REFERENCES:
- [Derived] Inoue Y, Hirata K, Hayashida K, Hattori N, Tomida T, Garcia-Borreguero D; Rotigotine Study Group. Efficacy, safety and risk of augmentation of rotigotine for treating restless legs syndrome. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Jan 10;40:326-33. doi: 10.1016/j.pnpbp.2012.10.012. Epub 2012 Oct 25. PMID 23103551

RESULTS

PARTICIPANT FLOW:
Groups:
- SPM 962: Rotigotine transdermal patch
  A patch containing 2.25 - 6.75mg of rotigotine was administered once a day.
Period: Overall Study
Arm/Group | SPM 962
Started | 185
Completed | 133
Not Completed | 52
Not completed — Adverse Event | 29
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 13
Not completed — Protocol Violation | 1
Not completed — Discontinuation criteria | 2
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | SPM 962
Number analyzed (Participants) | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 157
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 72
Region of Enrollment [Number; unit: participants]
  Japan | 185

OUTCOME MEASURES:

1. Primary Outcome: The Incidence and Severity of Adverse Events (AEs), Vital Signs, and Laboratory Parameters
Description: The safety of the long-term SPM 962 treatment was examined based on the incidence and severity of adverse events, vital signs, and laboratory parameters.
  AEs of special interest (1-3) are defined as below:
  1. sudden onset of sleep
  2. obsessive-compulsive disorder or impulse-control disorder
  3. hallucination, delusion
Time Frame: Up to 54 weeks
Population: Safety set (SS)
Measure: Number; unit: participants
Arm/Group | SPM 962
Number analyzed (Participants) | 185
participants
  Any AEs | 175
  Treatment-related AEs | 139
  SAEs | 5
  Treatment-related SAEs | 1
  Severe AEs | 3
  Discontinuation due to AEs | 29
  Death | 0
  AEs of special interest 1 | 0
  AEs of special interest 2 | 0
  AEs of special interest 3 | 0
  Valvular disease of the heart | 0

2. Primary Outcome: Augmentation
Description: Augmentation is the main complication during long-term dopaminergic treatment of restless legs syndrome (RLS) and reflects an overall increase in RLS severity.
  Augmentation is clinically significant when at least one of the following occurs:
  1. Change in daily activities and/or behavior (e.g., the patient stops riding in cars in the afternoon) due to augmentation;
  2. Negative impact on the patient's quality of life (sleep, mood, etc.) due to augmentation;
  3. Need to change the treatment dose or the patienｔ needs to take the dose earlier in the day (e.g., dividing the dose);
  4. Adjustments in concomitant medication are made to compensate for augmented RLS symptoms (e.g., an increased intake of analgesics or hypnotics to cover an increase in symptom intensity);
  5. Any other aspect as judged by the evaluator (should be specified).
Time Frame: Up to 53 weeks
Population: SS
Measure: Number; unit: participants
Arm/Group | SPM 962
Number analyzed (Participants) | 185
participants
  Subjects with augmentation | 11
  Subjects with clinically significant augmentation | 5

3. Secondary Outcome: Change of IRLS Sum Score From the Baseline to Each Visit
Description: IRLS is a scale for assessing severity of restless legs syndrome symptoms. IRLS consists of ten questions. Each question is scored from 4 for the first (top) answer (usually 'very severe') to 0 for the last answer (usually none).
  The sum of the score of each question serves as the scale score. The scale scoring criteria are: Mild (score 1-10); Moderate (score 11-20); Severe (score 21-30); Very severe (score 31-40). A decrease in the scores means improvement.
Time Frame: Baseline, Up to 53 weeks
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 184
Scores on a scale
  Weeks 8 | -11.4 (8.8)
  Week 16 | -9.7 (9.6)
  Week 32 | -9.5 (9.1)
  Week 44 | -10.4 (9.1)

4. Secondary Outcome: Efficacy Rate in IRLS Sum Score
Description: Efficacy rate (percentage of subjects with 50% decrease) (LOCF) in IRLS sum score.
Time Frame: Baseline, Up to 53 weeks
Population: FAS, LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SPM 962
Number analyzed (Participants) | 184
Percentage of participants
  Weeks 8 | 64.1 [57.2 to 71.1]
  Week 16 | 54.9 [47.7 to 62.1]
  Week 32 | 57.6 [50.5 to 64.7]
  Week 44 | 60.3 [53.3 to 67.4]

5. Secondary Outcome: Change of Augmentation Severity Rating Scale (ASRS) Sum Score From Baseline to Each Visit
Description: ASRS is a scale for assessing severity of augmentation. ASRS consists of 3 items (one item containing 4 sub-items). The sum of the score of each question serves as the scale score (each question score: 0-3, sum score 0-24).
  A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, Up to 52 weeks
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 184
Scores on a scale
  Week 8 | 1.4 (2.5)
  Week 16 | 1.4 (2.6)
  Week 32 | 1.6 (2.7)
  Week 44 | 1.4 (2.6)

6. Primary Outcome: Change of the Pittsburgh Sleep Quality Index (PSQI) From Baseline to Each Visit
Description: PSQI is a scale for assessing severity of sleep disorders. The score ranges from 0 to 21. 0 indicates "no difficulty" and 21 indicates "severe difficulty". A decrease in the scores means improvement.
Time Frame: Baseline, Up to 53 weeks
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 182
Scores on a scale
  Week 8 | -2.2 (3.3)
  Week 16 | -2.2 (2.9)
  Week 44 | -2.0 (3.1)

7. Secondary Outcome: Change of Short-Form 36-Item Health Survey (SF-36) From Baseline to Each Visit
Description: SF-36 is a scale for assessing health status in clinical practice and research. The scores of 36 questions are summarized into 7 sub-scales. In each sub-scale which range is 0-100, a higher score indicates a better health status. Thus a increase in the scores means improvement.
Time Frame: Baseline, Up to 53 weeks
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 182
Scores on a scale
  Physical functioning | -0.2 (8.0)
  Role physical | 3.7 (17.4)
  Bodily pain | 5.1 (22.3)
  General health | 1.8 (12.8)
  Vitality | 4.9 (15.8)
  Social functioning | 3.0 (16.2)
  Role emotional | 5.6 (14.5)

ADVERSE EVENTS:
Time Frame: 53 weeks
Arm/Group | SPM 962
Serious Adverse Events (participants affected / at risk) | 5/185
Other Adverse Events (participants affected / at risk) | 165/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=185)
Cataract (Eye disorders) | 1 (1)
Diverticulitis Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 (1)
Application Site Discolouration (General disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Neck Crushing (Injury, poisoning and procedural complications) | 1 (1)
Nerve Root Injury Lumbar (Injury, poisoning and procedural complications) | 1 (1)
Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=185)
Nausea (Gastrointestinal disorders) | 53 (79)
Vomiting (Gastrointestinal disorders) | 15 (26)
Diarrhoea (Gastrointestinal disorders) | 12 (12)
Abdominal Pain Upper (Gastrointestinal disorders) | 10 (11)
Application Site Reaction (General disorders) | 85 (94)
Application Site Pruritus (General disorders) | 12 (13)
Application Site Erythema (General disorders) | 6 (6)
Nasopharyngitis (Infections and infestations) | 97 (186)
Influenza (Infections and infestations) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 11 (11)
Contusion (Injury, poisoning and procedural complications) | 8 (8)
Blood Creatine Phosphokinase Increased (Investigations) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Headache (Nervous system disorders) | 25 (34)
Dizziness (Nervous system disorders) | 8 (12)
Somnolence (Psychiatric disorders) | 29 (33)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Eczema (Skin and subcutaneous tissue disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No